CLINICAL TRIAL: NCT03393208
Title: A Randomized, Open-label, 2-Way-Crossover Study Assessing the Bioequivalence Between Single Doses of 500 mg Glucophage Immediate Release (GIR) Tablets (Sino-American Shanghai Squibb Pharmaceuticals Ltd./ Manufactured in China) and 500 mg GIR Tablets (Merck Santé s.a.s. in Semoy/ Manufactured in France) Under Fed and Fasted State in Two Groups of Healthy Subjects
Brief Title: Glucophage Immediate Release (GIR) China Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200084_0009
Record Dates: First submitted 2017-12-22; First posted 2018-01-08 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Diabetes Mellitus; Glucophage Immediate Release (GIR); Bioequivalence Study
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First Test GIR (Fasting), Then Reference GIR (Fasting) (Experimental): Participants received a single oral dose of 500 milligram (mg) of test Glucophage Immediate Release (GIR) tablet Sino-American Shanghai Squibb (SASS)/China) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg reference GIR (Merck Santé in Semoy (MSS)/France) on Day 8 in treatment period 2 under fasting condition. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GIR; Drug: Reference GIR
- First Reference GIR (Fasting), Then Test GIR (Fasting) (Experimental): Participants received a single oral dose of 500 mg of reference GIR tablet (MSS/France) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg test GIR (SASS/China) on Day 8 in treatment period 2 under fasting condition. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GIR; Drug: Reference GIR
- First Test GIR (Fed), Then Reference GIR (Fed) (Experimental): Participants received a single oral dose of 500 mg of test GIR tablet (SASS/ China) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg reference GIR (MSS/France) on Day 8 in treatment period 2 under fed condition. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GIR; Drug: Reference GIR
- First Reference GIR (Fed), Then Test GIR (Fed) (Experimental): Participants received a single oral dose of 500 mg of reference GIR tablet (MSS/ France) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg test GIR (SASS/China) on Day 8 in treatment period 2 under fed condition. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GIR; Drug: Reference GIR

INTERVENTIONS:
Drug: Test GIR — Participants received 500 milligrams (mg) test GIR in fasting or fed state on either Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2).
  Other Names: Metformin
Drug: Reference GIR — Participants received 500 mg reference GIR in fasting or fed state on either Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2).
  Other Names: Metformin

SUMMARY:
The study will assess the bioequivalence between single doses of glucophage immediate release (GIR) test tablets and GIR reference tablets under fed and fasted state in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Participants had given written informed consent before any trial-related activities
* Chinese male and female participants (at least 1/4 of each gender per trial group)
* Aged between 18 and 55 years, inclusive
* Weighed: 50 to 80 kilogram (kg); Body mass index (BMI): 18 to 30 kg per meter square
* Nonsmoker since at least 3 months
* Good physical and mental health status, determined on the basis of the medical history and a physical examination
* All values for biochemistry and hematology tests of blood and urine within the normal range or showied no clinically relevant deviation as judged by the Investigator
* Electrocardiogram recording (12-lead ECG) without signs of clinically relevant pathology was judged by the Investigator
* Vital signs (blood pressure, pulse, body temperature, and respiration) in sitting position within the normal range or showing no clinically relevant deviation was judged by the Investigator
* All women of childbearing potential (WOCBP) who were not nursing, were not pregnant, and were using highly effective methods of birth control
* Negative screen for alcohol and drugs of abuse (cannabis, benzodiazepines, barbiturates, opiates, cocaine, and methyl amphetamine) were screened at and on admission
* Negative screen for hepatitis A virus (HAV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibodies, and Treponema pallidum (TP) antibodies

Exclusion Criteria:

* Participation in a clinical trial within 90 days prior to first drug administration
* Blood donation (equal or more than 500 milliliter [mL]) or significant blood loss within 90 days prior to first drug administration
* Any surgical or medical condition, including findings in the medical history or in the pretrial assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the participant in the trial or that could interfere with the trial objectives, conducted or evaluated
* History of surgery of the gastrointestinal tract which could influence the gastrointestinal absorption and/or motility according to the Investigator's opinion
* History or presence of relevant liver diseases or hepatic dysfunction Allergy: ascertained or presumptive hypersensitivity to the active drug substance and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considered affectted the outcome of the trial
* Receipt of any prescription or nonprescription medication within 2 weeks before the first IMP administration, including multivitamins and herbal products (example, St John's Wort, or traditional Chinese medicines), except paracetamol
* Renal failure or renal dysfunction (creatinine clearance < 80 mL/minute) as assessed by using the estimated measure with the Modification of Diet in Renal Disease (MDRD) equation
* Known lack of participant compliance or inability to communicate or cooperate with the Investigator (example, language problem and poor mental status)
* Nonacceptance of trial high-fat breakfast (example, vegetarians, vegans, and participants followed special diets)
* Consumption of large quantities of methyl xanthine-containing beverages (> 5 cups of coffee/day or equivalent)
* Consumption of grapefruit, cranberry or juices of these fruits, from 14 days prior to drug administration until collection of the last pharmacokinetic sample in Period 2
* Any contraindication to Glucophage
* Abnormal and clinically significant chest X-ray finding at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Xuanwu Hospital, Beijing, China

REFERENCES:
- [Derived] Hu C, Gao D, Li D, Zhou D, Zhang L. Chinese- and French-Manufactured Immediate-Release Glucophage(R) Bioequivalence: A Randomized, Open-Label, Crossover Study. Drugs R D. 2022 Dec;22(4):301-309. doi: 10.1007/s40268-022-00405-3. Epub 2022 Oct 20. PMID 36264446

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1 (Day 1-Day 3)
Arm/Group | First Test GIR (Fasting), Then Reference GIR (Fasting) | First Reference GIR (Fasting), Then Test GIR (Fasting) | First Test GIR (Fed), Then Reference GIR (Fed) | First Reference GIR (Fed), Then Test GIR (Fed)
Started | 13 | 13 | 9 | 9
Completed | 13 | 13 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Day 8- Day 10)
Arm/Group | First Test GIR (Fasting), Then Reference GIR (Fasting) | First Reference GIR (Fasting), Then Test GIR (Fasting) | First Test GIR (Fed), Then Reference GIR (Fed) | First Reference GIR (Fed), Then Test GIR (Fed)
Started | 13 | 13 | 9 | 9
Completed | 13 | 13 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Test GIR (Fasting), Then Reference GIR (Fasting) | First Reference GIR (Fasting), Then Test GIR (Fasting) | First Test GIR (Fed), Then Reference GIR (Fed) | First Reference GIR (Fed), Then Test GIR (Fed) | Total
Number analyzed (Participants) | 13 | 13 | 9 | 9 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (7.97) | 31.5 (7.39) | 29.8 (9.01) | 32.2 (7.03) | 31.7 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 4 | 14
  Male | 10 | 9 | 6 | 5 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 13 | 9 | 9 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-t) of Metformin (GIR Tablet Active Ingredient)
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 14 hours post-dose on Day 1; 24 and 36 hours post-dose on Day 2; 48 hours post-dose on Day 3
Population: The Pharmacokinetic (PK) Analysis Set included all participants who completed the study with adequate study drug compliance, without any relevant protocol violations with respect to factors likely to affect comparability of PK results, and with sufficient evaluable data to determine primary endpoints (AUC0-t and Cmax ) for both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Groups:
- Treatment A: Test GIR (Fasting): Participants received a single oral dose of 500 mg of test GIR tablet (SASS)/China) on Day 1 in treatment period 1 under fasting conditions.
- Treatment B Reference GIR (Fasting): Participants received a single oral dose of 500 mg of reference GIR tablet (MSS/ France) on Day 1 in treatment period 1 fasting conditions.
- Treatment A: Test GIR (Fed): Participants received a single oral dose of 500 mg of test GIR tablet (SASS/ China) on Day 8 in treatment period 2 under fed conditions.
- Treatment B: Reference GIR (Fed): Participants received a single oral dose of 500 mg of reference GIR tablet (MSS/ France) on Day 8 in treatment period 2 under fed conditions.
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 26 | 26 | 18 | 18
nanogram hour per milliliter (ng*h/mL) | 6260 (22.4) | 6280 (16.3) | 4950 (25.6) | 5020 (23.3)
Statistical Analysis 1: Comparison: Treatment A: Test GIR (Fasting) vs Treatment B Reference GIR (Fasting); Statistical Comparison of Treatment A Versus Treatment B in Fasting state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LeastSquare(LS) Mean% = 99.76, 90% CI 2-sided [92.84 to 107.20]
Statistical Analysis 2: Comparison: Treatment A: Test GIR (Fed) vs Treatment B: Reference GIR (Fed); Statistical Comparison of Treatment A Versus Treatment B in Fed state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 98.67, 90% CI [91.25 to 106.69]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metformin (GIR Tablet Active Ingredient)
Description: Pharmacokinetic (PK) parameter Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 26 | 26 | 18 | 18
ng/mL | 1110 (30.1) | 1110 (22.7) | 711 (22.4) | 700 (18.6)
Statistical Analysis 1: Comparison: Treatment A: Test GIR (Fasting) vs Treatment B Reference GIR (Fasting); Statistical Comparison of Treatment A Versus Treatment B in Fasting state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 99.62, 90% CI [92.69 to 106.77]
Statistical Analysis 2: Comparison: Treatment A: Test GIR (Fed) vs Treatment B: Reference GIR (Fed); Statistical Comparison of Treatment A Versus Treatment B in Fed state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 101.50, 90% CI [93.72 to 109.92]

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration of Metformin (GIR Tablet Active Ingredient)
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 26 | 26 | 18 | 18
hours | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.75 [1.50 to 5.00] | 2.75 [1.00 to 4.00]
Statistical Analysis 1: Comparison: Treatment A: Test GIR (Fasting) vs Treatment B Reference GIR (Fasting); Statistical Comparison of Treatment A Versus Treatment B in Fasting state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Median Difference = 0.00, 90% CI 2-sided [-0.25 to 0.25]
Statistical Analysis 2: Comparison: Treatment A: Test GIR (Fed) vs Treatment B: Reference GIR (Fed); Statistical Comparison of Treatment A Versus Treatment B in Fed state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Median Difference = 0.25, 90% CI [-0.25 to 0.50]

4. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Metformin (GIR Tablet Active Ingredient)
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set. Here "Number of particpants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 25 | 26 | 18 | 18
hours | 4.38 (40.5) | 4.90 (47.4) | 4.23 (45.6) | 4.16 (67.3)

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUCinf) of Metformin (GIR Tablet Active Ingredient)
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLQ) and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 25 | 26 | 18 | 18
ng*h/mL | 6520 (20.2) | 6410 (16.0) | 5070 (25.0) | 5160 (21.2)
Statistical Analysis 1: Comparison: Treatment A: Test GIR (Fasting) vs Treatment B Reference GIR (Fasting); Statistical Comparison of Treatment A Versus Treatment B in Fasting state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 101.26, 90% CI [94.33 to 108.69]
Statistical Analysis 2: Comparison: Treatment A: Test GIR (Fed) vs Treatment B: Reference GIR (Fed); Statistical Comparison of Treatment A Versus Treatment B in Fed state; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 98.17, 90% CI 2-sided [91.61 to 105.21]

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Tlast Extrapolated to Infinity (AUCextra) of Metformin (GIR Tablet Active Ingredient)
Description: AUCextra% was defined as area under the curve from time tlast extrapolated to infinity as percentage of AUC 0-infinity. Here, tlast is the last sampling time at which the concentration is at or above the lower limit of quantification.
Time Frame: as for outcome 1
Population: As AUCextra was >20% of AUC0-inf, parameters derived from λz including AUCextra% were regarded as unreliable estimate of the extent of exposure and not calculated.
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Elimination Rate Constant (λz) of Metformin (GIR Tablet Active Ingredient)
Description: λz was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 1
Population: As AUCextra was >20% of AUC0-inf, parameters derived from λz were regarded as unreliable estimate of the extent of exposure and not calculated.
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Total Body Clearance (CL/f) of Metformin (GIR Tablet Active Ingredient)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 25 | 26 | 18 | 18
liter per hour | 76.7 (20.2) | 78.0 (16.0) | 98.6 (25.0) | 96.8 (21.2)

9. Secondary Outcome: Apparent Volume of Distribution at After Extravascular Administration (Vz/f) of Metformin (GIR Tablet Active Ingredient)
Description: Vz/f is defined as the distribution of a study drug between plasma and the rest of the body after oral dosing.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set. . Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 25 | 26 | 18 | 18
liter | 485 (46.6) | 551 (52.5) | 602 (34.3) | 581 (73.1)

10. Secondary Outcome: Apparent Volume of Distribution at Steady-State After Extravascular Administration (Vss/f) of Metformin
Description: Vss/F was derived from concentration versus time data for all participants.
Time Frame: as for outcome 1
Population: As AUCextra was >20% of AUC0-inf, Vss/f derived from λz was regarded as unreliable estimate of the extent of exposure and not calculated.
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 15
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment B Reference GIR (Fasting: Participants received a single oral dose of 500 mg of reference GIR tablet (MSS/ France) on Day 1 in treatment period 1 fasting conditions.
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 26 | 26 | 18 | 18
Participants
  Any TEAE | 2 | 2 | 2 | 3
  Serious TEAE | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs, Laboratory Parameters, Physical Examination Findings and 12-lead Electrocardiogram (ECG) Findings
Description: The laboratory measurements included hematology, blood chemistry and urinalysis. Vital sign assessment included blood pressure, pulse rate and body temperature. ECG parameters included heart rate, PR, QRS,QT, RR, QTcB and QTcF Here, we are reporting number of participants with clinically significant abnormalities in Vital signs, laboratory parameters, physical findings and ECG findings.
Time Frame: Baseline up to Day 15
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug. Here "number of particpants were analyzed who were evaluable for this outcome measure".
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
Number analyzed (Participants) | 26 | 26 | 18 | 18
Participants
  Vital Signs | 0 | 0 | 0 | 0
  Laboratory Parameters | 0 | 0 | 0 | 0
  Physical Examination | 0 | 0 | 0 | 0
  12-Lead Electrocardiogram (ECG) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 15
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Treatment A Test GIR (Fasting): Participants received a single oral dose of 500 mg of test GIR tablet (SASS)/China) on Day 1 in treatment period 1 under fasting conditions.
Arm/Group | Treatment A Test GIR (Fasting) | Treatment B Reference GIR (Fasting) | Treatment A: Test GIR (Fed) | Treatment B: Reference GIR (Fed)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/26 | 2/26 | 2/18 | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A Test GIR (Fasting) (N=26) | Treatment B Reference GIR (Fasting) (N=26) | Treatment A: Test GIR (Fed) (N=18) | Treatment B: Reference GIR (Fed) (N=18)
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03393208/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03393208/SAP_001.pdf